CLINICAL TRIAL: NCT06389357
Title: Efficacy of the Web-based Return-to-school Adaptation Program for Children Diagnosed With Cancer
Brief Title: Retun-to-school Adaptation Program for Children With Cancer
Acronym: web-based
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gizem Çakır, Research Assistant, RN, PhD(c), Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1305G2024
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Childhood Cancer; ALL, Childhood; AML, Childhood; Lymphoma; Solid Tumor, Childhood
Keywords: childhood cancer; return to school; web-based programme; Got Transition; transition care; adaptation program; pediatric nursing; social anxiety; coping; readinness to return to school; Transition Theory
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma | interventions — Counseling; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: The research is a technical/scientific/collaborative action research design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implementation and evaluation of the school re-entry adaptation program (Experimental): Counselling interviews and workshops will be held simultaneously with the children receiving the web-based training. There are 4 modules in total. The first module lasts 2 weeks. The counselling interview will start in the 2nd week. Implementation will be completed in 5 weeks.
  Interventions: Behavioral: training and counselling; Other: Interview

INTERVENTIONS:
Behavioral: training and counselling — It includes 4 modules that develop children's communication, coping and social life skills and psychosocial preparation for the return to school process. The modules include theoretical explanations, stories, workshops and counselling sessions. Separate educational modules have been developed for parents, teachers, and peers.
  Other Names: workshops
Other: Interview — As part of the needs assessment in Phase 1, individual interviews with children with cancer and their parents lasting approximately 20-30 minutes were conducted.

SUMMARY:
The aim of this action research is to:

Stage 1: Conduct an in-depth investigation into the adaptation challenges faced by children aged 8-17 who are being treated for cancer during their return to school, from both the children's and parents' perspectives;

Stage 2: Develop a structured, evidence-based, and digitally accessible intervention program that addresses these identified needs;

Stage 3: Evaluate the feasibility and effectiveness of the intervention; and

Ultimately, based on all data gathered throughout the implementation process, continuously refine the intervention and analyze participant feedback holistically in order to establish a sustainable support model.

DETAILED DESCRIPTION:
Importance of research There are disease-specific medical and psychosocial difficulties that children with a diagnosis of cancer may experience. Standard school nursing practices can be helpful in meeting the physical, emotional, psychological, social and academic needs of children. However, a standard of care that is decided to be applied on return to school has not been developed. Therefore, it is thought that standard school nursing practices are not sufficient to meet the health and educational needs of children with cancer diagnosis. In the world, plans have been made using practices/methods/models appropriate for the population in the school return process of children followed up with a diagnosis of cancer. It is recommended to develop back-to-school programmes as they can benefit the child, family, peers, teachers and school staff who are followed up with a diagnosis of cancer. In our study, we aim to manage the transition care schematically with the back-to-school protocol to be made between the school-family-hospital, and to ensure care coordination and the safety of the child. The fact that the intervention in the back-to-school adaptation programme will be made to the child, parents, teachers and peers shows a holistic approach to the needs.

Place of application:

It will be performed in the paediatric leukaemia outpatient clinic of the Children's Hospital.

Study Population The population of the study consisted of children who were followed up in the paediatric leukaemia outpatient clinic of the Children's Hospital with a diagnosis of cancer.

Sample of the study In Phase 1, it was observed that after a certain number of interviews, no new themes or concepts emerged, and the data began to repeat previously obtained information. Accordingly, it was concluded that data saturation had been reached, and the data collection process was terminated. The sample for Phase 1 consisted of 12 children and their parents (n = 12).

In Phase 3, the study was conducted using a pre-experimental research design with a single group consisting only of the intervention group during the school re-entry adaptation program.

In program evaluation studies, a medium effect size is generally considered sufficient for quantitative evaluation methods. Accordingly, an effect size (Cohen's f) of at least 0.25 is recommended (Crisan & Elliott, 2018). For sample size planning, our study determined the estimated sample size to be 24 participants, based on 80% power and a 5% margin of error. The program in phase-3 was completed with 20 children and their parents who agreed to participate in the program.

Data Collection Tools

Phase 1: Identifying the experiences of children diagnosed with cancer and their parents during the return-to-school process - Descriptive phenomenological study:

The Child and Parent Descriptive Information Form Semi-Structured Interview Form

Phase 3: Implementation and evaluation of the school re-entry adaptation program:

1. Child and Parent Descriptive Information Form
2. Data Collection Form for Children's Return to School Process
3. Social Anxiety Scale for Children-Revised Version
4. Social Anxiety Scale for Adolescents
5. Paediatric Cancer Coping Scale
6. Readiness to Return to School Scale for Children with Oncological Problems: 7-18 Age
7. Process Evaluation Forms

Statistical analysis

Phase 1 - Qualitative Study:

The audio recordings of the interviews were transcribed. The qualitative data were analyzed using thematic content analysis via MAXQDA 2024 software. The steps of thematic analysis-transcription of the data, creation of codes, identification of themes, and reporting-were systematically followed to develop the context, main themes, and sub-themes. Codes were identified and grouped, which informed the final sub-theme and theme structure.

Sociodemographic characteristics collected during the qualitative phase were analyzed using SPSS version 30.0.0.0 and reported using frequencies and percentages.

Phase 3 - Implementation and Evaluation of the Program:

To assess the adaptation program, the normality of children's scale scores was evaluated using Shapiro-Wilk tests and skewness-kurtosis values. For variables that did not show a normal distribution, median values were reported (see Table 3.14).

The statistical significance of changes in scale scores over time within the sample group was examined using the Friedman test. A significance level of p ≤ 0.05 was accepted for all statistical tests. In cases where a statistically significant difference was found, Bonferroni-adjusted Wilcoxon Signed-Rank Tests were conducted to determine between which measurements the differences occurred, with a significance threshold set at p ≤ 0.01.

ELIGIBILITY:
Implementation and Evaluation of the School Re-entry Adaptation Program

Inclusion Criteria

For Children:

Aged between 8 and 17 years Diagnosed with cancer (leukemia, lymphoma, or solid tumor) For children diagnosed with leukemia, currently receiving or having completed maintenance therapy For children diagnosed with other cancer types, treatment has been completed or they are continuing outpatient treatment Have completed the treatment process but have not yet returned to school Have returned to school after treatment but discontinued again due to difficulties managing the adaptation process Have internet access Able to use the internet, computer, and phone Able to speak Turkish Consent to participate in the study

For Parents:

Own a computer or smartphone Have internet access Able to use the internet, computer, and phone Able to speak Turkish Consent to participate in the study

Exclusion Criteria

For Children:

Requiring special physical and/or mental care Having learning disabilities Having a psychological or medical diagnosis (e.g., severe depression) Diagnosed with brain tumor Diagnosed with osteosarcoma Receiving immunosuppressive therapy Experiencing a major stressful event within the past year (e.g., loss, surgery unrelated to cancer treatment) Preparing to take secondary or higher education entrance exams during the study period

For Parents:

Requiring special physical and/or mental care Having learning disabilities Having a psychological or medical diagnosis (e.g., severe depression)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
social anxiety | Before the intervention, before starting school, one month after starting school, three months after starting school
  Social anxiety scale fo children-revised. Scores that can be obtained from the scale are between 18-90 and as the scale score increases, the level of social anxiety increases.
coping | Before the intervention, before starting school, one month after starting school, three months after starting school
  Paediatric Cancer Coping Scale. Scores that can be obtained from the scale are between 0-99 and coping strategies increase as the scale score increases.
back to school readiness | Before the intervention, before starting school, one month after starting school, three months after starting school
  Back to school readiness scale for children with oncological problems: 7-18 years of age. The score that can be obtained from the scale is between 0 and 152 and a higher score indicates an increase in school readiness.

SECONDARY OUTCOMES:
process evaluation | 1st month and 3rd month after starting school
  Return to School Process Data Collection Form

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Cakir, PhD, Study Chair — Gazi University Nursing Faculty
Locations (1):
- Gizem Cakir, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared with other researchers. Since the data is individual, it is not ethically appropriate.

REFERENCES:
- [Background] Crisan A, Elliott M. How to evaluate an evaluation study? Comparing and contrasting practices in vis with those of other disciplines. IEEE Xplore. 2018; doi: 10.1109/BELIV.2018.8634420.
- [Background] Rabin C, Simpson N, Morrow K, Pinto B. Behavioral and psychosocial program needs of young adult cancer survivors. Qual Health Res. 2011 Jun;21(6):796-806. doi: 10.1177/1049732310380060. Epub 2010 Aug 12. PMID 20705863
- [Background] Ellis SJ, Wakefield CE, Antill G, Burns M, Patterson P. Supporting children facing a parent's cancer diagnosis: a systematic review of children's psychosocial needs and existing interventions. Eur J Cancer Care (Engl). 2017 Jan;26(1). doi: 10.1111/ecc.12432. Epub 2016 Jan 18. PMID 26776913
- [Background] Thompson AL, Christiansen HL, Elam M, Hoag J, Irwin MK, Pao M, Voll M, Noll RB, Kelly KP. Academic Continuity and School Reentry Support as a Standard of Care in Pediatric Oncology. Pediatr Blood Cancer. 2015 Dec;62 Suppl 5(Suppl 5):S805-17. doi: 10.1002/pbc.25760. PMID 26700927
- [Background] Canter KS, Roberts MC. A systematic and quantitative review of interventions to facilitate school reentry for children with chronic health conditions. J Pediatr Psychol. 2012 Nov-Dec;37(10):1065-75. doi: 10.1093/jpepsy/jss071. Epub 2012 Jun 19. PMID 22718487